CLINICAL TRIAL: NCT04333381
Title: Early Diagnosis of Acute Myocardial Infarction: Impact of an Educational and Organizational Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IIBSP-IAM-2015-84
Record Dates: First submitted 2020-03-24; First posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: STEMI; Myocardial Infarction; Nurses; Education; Emergency Room
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction; Emergencies

STUDY DESIGN:
Intervention Model Description: Quasi-experimental design study, pre-post intervention type
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Common Practice (Active Comparator): Patients included in the phase I will receive common practice.
  Interventions: Other: Common Practice
- Educational and organizational measures (Experimental): Patients included in the phase II will be attended by emergency nurses that received the educational and organizational intervention.
  Interventions: Other: Educational and organizational intervention

INTERVENTIONS:
Other: Educational and organizational intervention — Patients included after a systematic educational and organizational intervention for early diagnosis and care in myocardial infarction, aimed at emergency nurses of a tertiary Hospital capable in primary PCI.
  1. The educational intervention will consist:
     Systematized educational intervention on acute myocardial infarction for emergency triage nurses will consist of theoretical and practical training through case presentations and clinical simulation.
  2. The organizational intervention will consist:
     * Development and dissemination of an early diagnostic tool for acute myocardial infarction: STEMI infographics. It will be provided to all emergency nurses and emergency triage boxes
     * Update the STEMI hospital protocol and adapt it to the current clinical guidelines of the European Society of Cardiology (ESC)
     * Review organizational strategies and definition of new improvement measures
     * Audit the delays in STEMI
     * Periodic multi-disciplinary update sessions
  Arms: Educational and organizational measures
Other: Common Practice — Common practice is based on care by emergency nurses who did not receive any systematized education of acute myocardial infarction led by interventional cardiology nurses. On the other hand, emergency management is based on Plan-Do-Study-Act methodology and in the historical sample some organizational improvement strategies did not exist or were beginning to be implemented
  Arms: Common Practice

SUMMARY:
The hypothesis is that an educational program aimed at emergency nurses and the implementation of measures at the organizational level reduce the time between arrival at the emergency room and the opening of the artery or balloon by 40% in patients attending for acute myocardial infarction.

DETAILED DESCRIPTION:
The time between arrival in the emergency room (ER) and balloon time (D2B) in ST segment elevation myocardial infarction (STEMI) is one of the best indicators of quality care in patients with STEMI. Hospitals with more strategies to improve this quality of care have a shorter door-to-balloon time. The aim is to evaluate the effectiveness, in the time between the arrival in the ER and the balloon time, of an educational and organizational intervention for the early diagnosis of myocardial infarction for emergency nurses.

The aim of this study is to improve the time between arrival to ER and balloon time.

The study consists of two phases:

Phase I (PRE): in this phase, the aim is to describe the attendance times and to evaluate the causes of delay in attendance in STEMI patients. With the findings, a plan will be drawn up that includes the integration of an educational program for emergency nurses and organizational measures; oriented to improve the early diagnosis and delays in STEMI.

Phase II (POST): in this phase, the aim is to evaluate the effectiveness in improving delays in the care of patients with STEMI after the implementation of the educational and organizational intervention developed in phase 1. On the other hand, will evaluate the satisfaction of the emergency nurses with the training they received through educational and organizational intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years
* Admitted to the emergency room of the same center

Exclusion Criteria:

* Pregnant women
* Patients who did not receive coronariography were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Door-to-balloon time (D2B) | up to 30 days; From the arrival at the emergency room to the balloon time up to discharge
  The time between arrival at the emergency room (ER) and balloon time (D2B) in STEMI

SECONDARY OUTCOMES:
ER arrival-ECG time | up to 30 days; from the arrival at the emergency department to the ECG realization up to discharge
  The time between the arrival at the emergency department and the ECG.

CONTACTS AND LOCATIONS:
Locations (1):
- FGS Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

REFERENCES:
- [Derived] Berga Congost G, Martinez Momblan MA, Valverde Bernal J, Marquez Lopez A, Ruiz Gabalda J, Garcia-Picart J, Puig Campmany M, Brugaletta S. Association of sex and age and delay predictors on the time of primary angioplasty activation for myocardial infarction patients in an emergency department. Heart Lung. 2023 Mar-Apr;58:6-12. doi: 10.1016/j.hrtlng.2022.10.014. Epub 2022 Nov 3. PMID 36335910
- [Derived] Berga Congost G, Brugaletta S, Valverde Bernal J, Marquez Lopez A, Ruiz Gabalda J, Garcia-Picart J, Puig Campmany M, Martinez Momblan MA. The importance of organizational variables in treatment time for patients with ST-elevation acute myocardial infarction improve delays in STEMI. Australas Emerg Care. 2021 Jun;24(2):141-146. doi: 10.1016/j.auec.2020.10.001. Epub 2020 Nov 14. PMID 33199195